CLINICAL TRIAL: NCT04350801
Title: Usefulness of a Home-based Cognitive Monitoring in Non-demented Patients With High-risk of Dementia: a Prospective Observational Study
Brief Title: Home-based Cognitive Monitoring in MCI
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Asan Medical Center (Other)
Responsible Party: Principal Investigator, YunJeong Hong, MD, professor, Asan Medical Center
Other Study IDs: Hom-based cognitive monitoring
Record Dates: First submitted 2020-04-15; First posted 2020-04-17 (Actual); Last update posted 2020-04-20 (Actual); Status verified 2020-04

CONDITIONS: Mild Cognitive Impairment
Keywords: mild cognitive impairment; blood amyloid beta; home-based cognitive monitoring
MeSH Terms: conditions — Cognitive Dysfunction

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- high risk MCI: MCI patients with amyloid beta positive (based on peripheral blood level)
  Interventions: Diagnostic Test: home-based cognitive monitoring
- low risk MCI: MCI patients with amyloid beta negative (based on peripheral blood level)
  Interventions: Diagnostic Test: home-based cognitive monitoring

INTERVENTIONS:
Diagnostic Test: home-based cognitive monitoring — a newly developed home-based cognitive monitoring (about 3-5 minutes per test; total score ranges from 0~30; higher score indicates better cognition)

SUMMARY:
This study is an observational study to confirm usefulness of a home-based cognitive monitoring in non-demented patients with high-risk of dementia

DETAILED DESCRIPTION:
We prospectively enroll subjects who were diagnosed as mild cognitive impairment based on neuropsychological tests battery, brain MRI, and routine blood labs including thyroid function tests, vitamine B12 & folate levels, and syphilis screening to rule out other secondary causes of dementia. We undergo peripheral blood-based amyloid beta levels and regular home-based cognitive monitoring (every 3 months) to investigate whether amyloid-positive MCIs progress rapidly using home-based cognitive monitoring during 6 months.

ELIGIBILITY:
Inclusion Criteria:

* persistent cognitive complaints
* aged 50 years old or older
* below -1.0 standard deviation in any domain of detailed neuropsychological tests battery named SNSB (Seoul neuropsychological screening battery)
* no ADL (activities of daily living) limitation
* subjects who agreed to participate

Exclusion Criteria:

* dementia patients
* other structural brain disorders such as hydrocephalus, hemorrhage, or tumors
* other neurological disease such as Huntington's disease, Parkinson's disease, or epilepsy

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: clinically diagnosed mild cognitive impairment according to Petersen's criteria
Sampling Method: Probability Sample
Enrollment: 40 (Estimated)
Dates: Start 2019-12-01 (Actual); Primary Completion 2020-11-01 (Estimated); Study Completion 2020-12-30 (Estimated)

PRIMARY OUTCOMES:
home-based cognitive monitoring score | 3 months (at baseline, 3 months from baseline, 6 months from baseline)
  a 3-5 minutes brief cognitive testing (range 0~30, higher score means better outcome) using telephone

SECONDARY OUTCOMES:
Hippocampal atrophy grade | at baseline
  baseline brain MRI markers for hippocampal atrophy using Scheltens' visual rating scale (range 0~4, higher score means more hippocampal atrophy)
Number of lacunes | at baseline
  number of lacunes using manual counting on brain MRI (no limit)
Number of microbleeds | at baseline
  number of microbleeds using manual counting on brain MRI (no limit)

CONTACTS AND LOCATIONS:
Overall Officials: YunJeong Hong, MD, PhD, Principal Investigator — Uijeongbu St. Mary's Hospital
Locations (1):
- Uijeongbu St. Mary's hospital, Uijeongbu-si, South Korea

IPD SHARING:
Plan to Share IPD: No